CLINICAL TRIAL: NCT07042919
Title: A Phase Ib/II Study of Zanzalintinib in Second Line and Beyond for the Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Zanzalintinib in Second Line and Beyond for the Treatment of Advanced Liver Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 25I02; NCI-2025-04131 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00223939; NU 25I02 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Advanced Hepatocellular Carcinoma; Cirrhosis; Stage III Hepatocellular Carcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular | interventions — Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (zanzalintinib) (Experimental): Patients receive zanzalintinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA at baseline and urine and blood sample collection and CT or MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Zanzalintinib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo urine and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Zanzalintinib — Given PO
  Other Names: Multi-kinase Inhibitor XL092; XL 092; XL-092; XL092

SUMMARY:
This phase Ib/II trial tests the safety, side effects, and best dose of zanzalintinib and how well it works in treating patients with hepatocellular (liver) cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). Zanzalintinib is in a class of medications called tyrosine kinase inhibitors. It works by blocking the action of an abnormal protein that signals tumor cells to multiply, which may help keep tumor cells from growing. Giving zanzalintinib may be safe, tolerable, and/or effective in treating patients with advanced liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety, tolerability, and dose limiting toxicity (DLT) in patients with advanced hepatocellular carcinoma (aHCC, Child-Pugh class A and B cirrhosis) and the determination of the recommended phase II dose (RP2D) with zanzalintinib. (Phase Ib dose escalation only)

SECONDARY OBJECTIVES:

I. Assess the proportion of aHCC zanzalintinib treated patients that are alive and median progression-free survival (PFS) of treatment. (Phase Ib and Phase II) II. Assess median overall survival (OS) in aHCC zanzalintinib treated patients. (Phase Ib and Phase II) III. Assess the proportion of aHCC zanzalintinib treated patients that have an objective response to treatment by imaging.

EXPLORATORY (CORRELATIVE) OBJECTIVE:

I. Assess correlatives and the pharmacokinetics (PK) profile by biomarker assessment during treatment of aHCC patients with zanzalintinib.

OUTLINE: This is a phase Ib dose-escalation study followed by a phase II dose-expansion study.

Patients receive zanzalintinib orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) at baseline and urine and blood sample collection and computed tomography (CT) or magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosed hepatocellular carcinoma (HCC) who are not amendable to curative treatments
* Patients must have documented objective radiographic progression during or after treatment with any first or second line therapy, or intolerance to any first or second line therapy, which include immunotherapy-based combination, or non-immunotherapy-based treatment, except cabozantinib
* Patients must have a Child-Pugh class A or Child-Pugh class B (B7 or B8) score for cirrhosis mortality. Child-Pugh class B, B9 is excluded
* Patients must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
* Patients may have had up to two prior lines therapy (not including cabozantinib) in the advanced metastatic setting. Palliative radiation or locoregional therapies are not considered a line of therapy
* Patients must be age ≥ 18 years
* Patients must exhibit a/an Eastern Cooperative Oncology Group (ECOG) Status of 0-1 (Karnofsky ≥ 60%)
* CHILD-PUGH CLASS A: Absolute neutrophil count (ANC) ≥ 1,500/mcL without granulocyte colony-stimulating factor support within 2 weeks of screening laboratory sample collection
* CHILD-PUGH CLASS B: Absolute neutrophil count (ANC) ≥ 1,200/mcL without granulocyte colony-stimulating factor support within 2 weeks of screening laboratory sample collection
* CHILD-PUGH CLASS A: Hemoglobin (Hgb) ≥ 9 g/dL without transfusion within 2 weeks of screening laboratory sample collection
* CHILD-PUGH CLASS B: Hemoglobin (Hgb) ≥ 8.5 g/dL without transfusion within 2 weeks of screening laboratory sample collection
* CHILD-PUGH CLASS A: Platelets (PLT) ≥ 75,000/mcL without transfusion within 2 weeks of screening laboratory sample collection
* CHILD-PUGH CLASS B: Platelets (PLT) ≥ 60,000/mcL without transfusion within 2 weeks of screening laboratory sample collection
* CHILD-PUGH CLASS A: International normalized ratio (INR) ≤ 1.7 x upper limit of normal (ULN)
* CHILD-PUGH CLASS B: International normalized ratio (INR) ≤ 2.3 x upper limit of normal (ULN)
* CHILD-PUGH CLASS A: Activated partial thromboplastin time (aPTT) ≤ 1.2 x upper limit of normal (ULN)
* CHILD-PUGH CLASS B: Activated partial thromboplastin time (aPTT) ≤ 1.2 x upper limit of normal (ULN)
* CHILD-PUGH CLASS A: Total bilirubin ≤ 3.0 mg/dl (For subjects with Gilbert's disease ≤ 3 x ULN)
* CHILD-PUGH CLASS B: Total bilirubin ≤ 3.0 mg/dl (For subjects with Gilbert's disease ≤ 3 x ULN)
* CHILD-PUGH CLASS A: Albumin ≥ 2.5 (g/dL)
* CHILD-PUGH CLASS B: Albumin ≥ 2.5 (g/dL)
* CHILD-PUGH CLASS A: Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) ≤ 5 x institutional ULN (specify modifications for liver metastases, as applicable)
* CHILD-PUGH CLASS B: AST (SGOT) ≤ 5 x institutional ULN (specify modifications for liver metastases, as applicable)
* CHILD-PUGH CLASS A: Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 5 x institutional ULN (specify modifications for liver metastases, as applicable)
* CHILD-PUGH CLASS B: ALT (SGPT) ≤ 5 x institutional ULN (specify modifications for liver metastases, as applicable)
* CHILD-PUGH CLASS A: Alkaline phosphatase (ALP) ≤ 5.0 x institutional ULN
* CHILD-PUGH CLASS B: ALP ≤ 5.0 x institutional ULN
* CHILD-PUGH CLASS A: Creatinine clearance > 40 mL/ minute if serum creatinine is elevated above 1.5 x ULN
* CHILD-PUGH CLASS B: Creatinine clearance > 40 mL/ minute if serum creatinine is elevated above 1.5 x ULN
* CHILD-PUGH CLASS A: Urine protein-to-creatinine ratio (UPCR) ≤ 1.5 mg/mg (≤ 169.8 mg/mmol) creatinine
* CHILD-PUGH CLASS B: Urine protein-to-creatinine ratio (UPCR) ≤ 1.5 mg/mg (≤ 169.8 mg/mmol) creatinine
* Patients of child-bearing potential (POCBP) and any of their partners with sperm-producing reproductive capability must agree to use a highly effective method of contraception throughout the course of the study and for 186 days after the last dose of treatment. Additional contraceptive method, such as a barrier method (e.g., condom) is also required
* Patients with sperm-producing reproductive capacity (PWSPRC) treated or enrolled on this protocol must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) with partners of childbearing potential from time of informed consent, for the duration of study participation, and for 96 days following completion of therapy
* POCBP must agree to use a highly effective method of contraception throughout the course of the study and for 186 days after the last dose of treatment. Additional contraceptive method, such as a barrier method (e.g., condom) is also required
* Patients must have the ability to understand and the willingness to sign a written informed consent document and comply with the study requirements
* Patients must have the ability to swallow, retain, and absorb oral medications or ingest a suspension either orally or by a nasogastric (NG) or gastrostomy (PEG) tube

Exclusion Criteria:

* Patients with prior treatment with zanzalintinib
* Patients who have received any type of small-molecule kinase inhibitor (including an investigational kinase inhibitor) within 14 days prior to study day 1 treatment
* Patients who have received ≥ 3 prior therapies in the advanced setting
* Patients with prior Cabozantinib use
* Patients who have had chemotherapy, cytotoxic, biologic, radiation, or other systemic anticancer (including investigational) therapy within 4 weeks prior to study day 1 treatment
* Patients who have received palliative radiation therapy for bone metastasis within 14 days or any other radiation therapy within 4 weeks days before first dose of study treatment
* Patients who have undergone systemic treatment with radionuclides within 6 weeks (42 days) before first dose of study treatment
* Patients who have received any local anticancer therapy including surgery, percutaneous ethanol injection (PEI), radiofrequency ablation (RFA), microwave ablation (MWA), transarterial chemoembolization (TACE), or trans arterial radioembolization (TARE) within 28 days prior to first dose of study treatment
* Patients with any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE 5.0) grade > 1 at baseline, including immune-related adverse events (irAEs), related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy (eg, physiological replacement of corticosteroid, from a previous anticancer therapy, with the following exceptions:

  * Alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
  * Patients with grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the treating physician
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with zanzalintinib may be included only after consultation with the principal investigator
* Patients with a known prior or concurrent malignancy that is progressing or requires active treatment within 2 years of first dose of study treatment

  * Note: The following exceptions may be made:

    * For patients with malignancies like basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer; or superficial skin cancers, localized low-grade tumors deemed cured and not treated with systemic therapy, and incidentally diagnosed prostate cancer if assessed as stage ≤ T2N0M0 and Gleason score ≤ 6
    * For patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Patients with known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 28 days prior to first dose of study treatment

  * Note: Patients with an incidental finding of an isolated brain lesion < 1 cm in diameter may be eligible after principal investigator approval if the lesion is radiographically stable for 28 days before first dose and does not require treatment per Investigator judgement
  * Note: Eligible patients must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment
  * Note: Base of skull lesions without definitive evidence of dural or brain parenchymal involvement are allowed
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to zanzalintinib
* Patients who are on concomitant anticoagulation therapy with oral anticoagulants (e.g., warfarin or direct thrombin inhibitors) and platelet inhibitors (e.g., clopidogrel)

  * Allowed anticoagulants are the following:

    * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH)
    * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in patients without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen
  * Note: Patients must have discontinued oral anticoagulants within 3 days or 5 half-lives prior to first dose of study treatment, whichever is longer
* Patients who are taking any complementary medications (e.g., herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks prior to cycle 1 day 1

  * Note: Taking complementary medications to treat symptoms of the cancer is allowed
* Patient has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Deteriorating Cardiovascular disorders:

    * Congestive heart failure (CHF) New York Heart Association class 3 or 4, class 2 or higher unstable angina pectoris, new-onset angina, serious cardiac arrhythmias (e.g., ventricular flutter, ventricular fibrillation, Torsades de pointes)
    * Ejection fraction < 50% on screening echocardiogram (ECHO) or multigated acquisition scan (MUGA)
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic of > 90 mm Hg diastolic despite optimal antihypertensive treatment
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction, or other clinically significant ischemic events within 6 months prior to first dose of study treatment
    * Pulmonary embolism (PE) or deep vein thrombosis (DVT) or prior clinically significant venous or non-CVA/TIA arterial thromboembolic events within 3 months before to first dose of study treatment

      * Note: Patients with a diagnosis of DVT within 6 months are allowed if asymptomatic and stable at screening and are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen
      * Note: Patients who don't require prior anticoagulation therapy may be eligible but must be discussed and approved by the principal investigator
    * Prior history of myocarditis
  * Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

    * Tumors invading the GI tract from external viscera
    * Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis
    * Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess must be confirmed prior to first dose of study treatment
    * Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment
    * Known gastric or esophageal varices
    * Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months unless cause of obstruction is definitively managed and patient is asymptomatic
* Patients with clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 mL) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 84 days prior to registration
* Patients with symptomatic cavitating pulmonary lesion(s) or endobronchial disease (asymptomatic or radiated lesions allowed)
* Patients with lesions invading major blood vessel including but not limited to inferior vena cava, pulmonary artery, or aorta

  * Note: Patients with intravascular tumor extension (e.g., tumor thrombus in renal vein or inferior vena cava) may be eligible following principal investigator (PI) approval. Patients with lesions invading the hepatic portal vasculature are eligible
* Patients with other clinically significant disorders that would preclude safe study participation, including, but not limited to:

  * Active infection requiring systemic treatment

    * Note: This criterion applies only at enrollment; if a patient develops an infection while on study treatment, they may continue to receive study treatment
    * Note: prophylactic antibiotic treatment is allowed
  * Known infection with acute hepatitis B virus (HBV)

    * Note: Subjects with active hepatitis B virus (HBV) infection (defined by hepatitis B virus surface antigen [HBsAg] positive) must be on standard of care antiviral therapy and have HBV deoxyribonucleic acid (DNA) < 500 IU/mL. Please note this lab is not a requirement for eligibility, however if it has been completed previously as part of the patient's health care, it should be documented for eligibility
  * Patients with active, uncontrolled hepatitis C virus infection are eligible provided liver function meets eligibility criteria and are receiving management of the disease per local institutional practice

    * Note: antiviral treatment for hepatitis C virus (HCV) is allowed with PI approval
  * Known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness

    * Note: except for patients meeting all of the following criteria:

      * On stable anti-retroviral therapy
      * CD4+ T cell count ≥ 200/uL
      * An undetectable viral load
    * Note: To be eligible, participants taking cytochrome P450 (CYP) inhibitors (eg, zidovudine, ritonavir, cobicistat, didanosine) or CYP3 inducers (efavirenz) must change to a different regimen not including these drugs 7 days prior to initiation of study treatment. Anti-retroviral therapies (ART) must have been received for at least 28 days prior to the first dose
    * Note: CD4+ T cell counts, and viral load are monitored per standard of care by the local health care provider
  * Serious non-healing wound/ulcer/bone fracture

    * Note: non-healing wounds or ulcers are permitted if they are due to tumor-associated skin lesions
  * Malabsorption syndrome
  * Pharmacologically uncompensated, symptomatic hypothyroidism
  * Severe hepatic impairment (Child-Pugh C)
  * Requirement for hemodialysis or peritoneal dialysis
  * History of solid organ or allogeneic stem cell transplant
* Patients with Recent surgery within the following parameters:

  * Major surgery (e.g., GI surgery or removal/biopsy of brain metastasis) within 8 weeks before first dose of study treatment
  * Prior laparoscopic surgeries (i.e. nephrectomy) within 28 days prior to first dose of study treatment. Minor surgery (e.g., simple excision, tooth extraction) within 5 days before first dose of study treatment
  * Complete wound healing from major surgery and from minor surgery (e.g., simple excision, tooth extraction) must have occurred at least prior to first dose of study treatment
  * Patients with clinically relevant ongoing complications from prior surgery are not eligible
  * Minor surgery (e.g., simple excision, tooth extraction) within 5 days prior to first dose of study treatment

    * Note: if a patient has had a recent surgery outside of the proscribed interval, complete wound healing from said surgery must have occurred prior to first dose of study treatment
    * Note: Fresh tumor biopsies should be performed at least 5 days prior to registration. Patients with clinically relevant ongoing complications from prior surgical procedures, including biopsies, are not eligible
* Patients with corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms within 14 days per electrocardiogram (ECG) prior to first dose of study treatment

  * Note: Triplicate ECG evaluations will be performed and the average of these 3 consecutive results for QTcF will be used to determine eligibility
* Patients who are pregnant (positive serum or urine test within 72 hours prior to enrollment) or nursing. Pregnant people are excluded from this study because zanzalintinib is a next-generation tyrosine kinase inhibitor (TKI) with potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the nursing parent with zanzalintinib , breastfeeding should be discontinued if the nursing parent is treated with zanzalintinib

  * POCBP are considered to be of childbearing potential unless one of the following criteria is met: permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, POCBP < 55 years-of-age must have a serum follicle stimulating hormone [FSH] level > 40 mIU/mL to confirm menopause)
  * Note: Documentation may include review of medical records, medical examination, or medical history interview by study site staff
  * Note: If a urine pregnancy test is positive or cannot be confirmed negative, a serum pregnancy test will be required
* Patients with psychiatric illness/social situations that would limit compliance with study requirements or give informed consent, per the opinion of the treating investigator
* Patients with other conditions which, in the opinion of the investigator, would compromise the safety of the patient or the patient's ability to complete the study
* Patients with documented hepatic encephalopathy (HE) within 6 weeks before first dose of study treatment

  * Patients with clinically meaningful ascites (i.e., ascites requiring paracentesis or escalation in diuretics) within 2 weeks prior to registration, cycle 1 day 1 (C1D1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2026-03-04 (Estimated); Primary Completion 2029-03-04 (Estimated); Study Completion 2031-03-04 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) (Phase Ib dose-escalation only) | Through the duration of cycle 1 (cycle length = 28 days)
  Will be reported using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Will be sorted by type, severity (grade), timing and attribution to zanzalintinib. Will be evaluated using descriptive statistics to summarize the frequency and severity. The number and proportion of patients experiencing DLTs will be reported, with each patient counted only once, regardless of the number of DLTs experienced.
Recommended phase 2 dose (Phase Ib dose escalation only) | Up to 1 year
  Will be defined as the dose level that does not exceed the DLT limit established by the dose escalation plan per cohort.
Incidence of adverse events (AEs) (Phase Ib) | Up to 30 days from last dose of study treatment
  AEs and serious AEs will be reported using CTCAE v 5.0. Will be sorted by type, severity (grade), timing and attribution to zanzalintinib. The frequency of treatment discontinuations due to toxicity will also be reported. These data will be presented using descriptive statistics, including counts and percentages for categorical variables, and means or medians with standard deviations or interquartile ranges for continuous variables.

SECONDARY OUTCOMES:
Incidence of AEs | Up to 30 days after last dose of study treatment
  AEs and serious AEs will be reported using CTCAE v 5.0. Will be sorted by type, severity (grade), timing and attribution to zanzalintinib.
Median progression-free survival (PFS) (Phase Ib and II) | From start of trial therapy (cycle 1 day 1 [cycle length = 28 days]) until disease progression, initiation of subsequent anti-cancer therapy, study completion, or death from any cause, whichever occurs first, assessed up to 1 year
  Will be determined by radiographic imaging as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 criteria. Will be analyzed using Kaplan-Meier survival analysis. Kaplan-Meier curves will be generated to estimate PFS rates at the specified time points, and median PFS will be reported along with 95% confidence intervals. Additionally, Cox proportional hazards regression models may be used to adjust for potential confounders and to estimate hazard ratios for progression or death.
Overall survival (Phase Ib and II) | From the start of trial therapy to the time of death from any cause, assessed up to 1 year
Objective response rate | Up to 1 year
  Will be defined as the proportion of treated subjects who experience confirmed complete response or confirmed partial response per RECIST v 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Devalingam Mahalingam, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States